CLINICAL TRIAL: NCT03705780
Title: Comparison of Preoperative Fentanyl Test and A Short OSAS Screening Scale for Identifying Severe Obstructive Sleep Apnea Syndrome
Brief Title: Fentanyl Test and A Short OSAS Screening Scale for Severe Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Xuan Wang, Director，Head of Anesthesiology, Children's Hospital of Fudan University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: FTASOSSSOSP
Record Dates: First submitted 2018-09-25; First posted 2018-10-15 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: fentanyl; OSAS screening scale; adenotonsillectomy; diagnose
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the short OSAS scale (Other): In preoperative interview，distributing the short OSAS screening scales to children's parents，and the scale was completed preoperative，calculate the score of the scale
  Interventions: Other: the short OSAS scale
- fentanyl test (Experimental): In the operating room，giving 1 mcg/kg fentanyl when the End-tidal concentrations of sevoflurane were maintained at 3.0 and the spontaneous respiratory frequency was stable after eyelash reflex disappeared and pharyngeal airway insertion, observing the changes of respiratory rate
  Interventions: Diagnostic Test: fentanyl test

INTERVENTIONS:
Other: the short OSAS scale — Parents fill in the short OSAS screening scale in preoperative interview，calculate score of the scale.
  Arms: the short OSAS scale
Diagnostic Test: fentanyl test — In the operating room，giving 1 mcg/kg fentanyl when the End-tidal concentrations of sevoflurane were maintained at 3.0 and the spontaneous respiratory frequency was stable after eyelash reflex disappeared and pharyngeal airway insertion, observing the changes of respiratory rate
  Arms: fentanyl test

SUMMARY:
The aim of this study was to estimate and compare the value of the preoperative fentanyl test and the short OSAS screening scale to diagnose severe obstructive sleep apnea；and to observe the required amount of hydromorphone and the adverse respiratory events after adenotonsillectomy.

DETAILED DESCRIPTION:
The results of polysomnography were obtained before adenotonsillectomy, and the short OSAS screening scale was completed by the subjects' parents in preoperative interview. All children were induced by sevoflurane inhalation. After eyelash reflex disappeared and pharyngeal airway insertion, giving 1 mcg/kg fentanyl when the End-tidal concentrations of sevoflurane were maintained at 3.0 and the spontaneous respiratory frequency was stable, observing the changes of respiratory rate. Severe OSAS was diagnosed as respiratory rate decreased by more than 50%. Anesthesia was maintained with desflurane and 60% nitrous oxide in oxygen. The children were transferred to the PACU after extubation. The postoperative pain and agitation were assessed according to the Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) and The Pediatric Anesthesia Emergency Delirium (PAED) score, and all children were given hydromorphone for pain relief according to our protocol.

ELIGIBILITY:
Inclusion Criteria:

1. The American society of anesthesiologists (ASA) class Ⅰ ~ Ⅱ
2. Age greater than or equal to 3 years
3. Children were diagnosed by polysomnography and plan to adenotonsillectomy.

Exclusion Criteria:

1. craniofacial malformations
2. mental retardation
3. BMI > 30 kg/m2
4. Combined with other neuromuscular diseases
5. a recent history of opioid use

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity， specificity ，positive predictive value and negative predictive value，likelihood ratio | 5 months
  Compared the diagnostic results of fentanyl test and the short OSAS screening scale with the diagnostic results of golden standard PSG.

SECONDARY OUTCOMES:
hydromorphone requirement in PACU | 50 minutes after extubation
  Pain was assessed according to the Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) and hydromorphone of 2 µg/Kg was provided if the CHEOPS pain score was >6.
  The CHEOPS is a behavioral scale for evaluating postoperative pain in young children. It can be used to monitor the effectiveness of interventions for reducing the pain and discomfort.It includes six categories of pain behavior, each with 3-4 levels.
  CHEOPS pain score = SUM(points for all 6 parameters)
  minimum score: 4 maximum score: 13

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Wang, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Chilren's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No